CLINICAL TRIAL: NCT06767228
Title: The Effects of Reformer Pilates Exercises on Trunk Endurance, Posture, and Body Awareness in Adolescents
Brief Title: Effects of Reformer Pilates on Adolescents' Posture and Trunk Endurance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Muhammed Şeref Yıldırım, Research Assistant (PhD), Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TU-FTR-MŞY-003
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Adolescent; Healthy
Keywords: Adolescent; Exercise therapy; Posture; Body awareness

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two parallel groups: one receiving reformer pilates exercises and the other receiving educational sessions on posture and physical activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reformer Pilates Group (Experimental): Participants in this group will perform reformer pilates exercises twice weekly for six weeks. Each session will last 50 minutes and include warm-up, main exercises, and cool-down phases.
  The exercises will target both deep and superficial core muscles, focusing on core endurance, posture, and body awareness.
  The main program includes 12 reformer exercises (e.g., Footwork Series, Pelvic Lift, Arm Circles, Leg Circles) with progressive resistance and repetitions (10 repetitions for the first 3 weeks and 15 repetitions for the last 3 weeks).
  The intervention will be carried out under professional supervision. Cool-down includes diaphragmatic breathing and relaxation-focused Footwork exercises.
  Interventions: Behavioral: Reformer Pilates
- Educational Session Group (No Intervention): Participants in this group will receive a one-time, 60-minute educational session on proper posture and the importance of physical activity at the start of the study. This session will include:
  Verbal and visual explanations about maintaining correct postural alignment in daily activities such as sitting, standing, and lifting.
  Practical tips on integrating physical activity into their daily routines to support overall health and posture.
  No structured exercise or physical activity will be performed during the six-week study period. Participants will be invited to post-intervention assessments after six weeks. Additionally, participants will be offered the opportunity to join the reformer pilates exercise program after the study concludes, if they wish.

INTERVENTIONS:
Behavioral: Reformer Pilates — This intervention involves a structured reformer pilates program designed to enhance core endurance, posture, and body awareness. The program includes exercises such as Footwork Series, Pelvic Lift, Arm Circles, Leg Circles, Frog Series, Long Box Series, Short Box Series, Elephant, Knee Stretch Series, Stomach Massage, and Side Stretch. The program emphasizes progressive resistance, controlled movements, and professional supervision to ensure safety and effectiveness. Sessions are conducted twice weekly for six weeks.
  Arms: Reformer Pilates Group

SUMMARY:
This study aims to investigate the effects of reformer pilates exercises on posture, core endurance, and body awareness in adolescents. The hypothesis is that reformer pilates will improve these outcomes compared to a control group receiving only informational support. Participants will be randomized into two groups and assessed over six weeks.

DETAILED DESCRIPTION:
This randomized controlled trial investigates the effects of reformer pilates exercises on core endurance, posture, and body awareness in adolescents aged 10-19. Participants will be randomly assigned to one of two groups: an intervention group performing reformer pilates exercises and a control group receiving educational information on posture and physical activity. Both groups will be assessed at baseline and after the 6-week intervention period.

A. Study Design

Intervention Group: Participants in this group will perform reformer pilates exercises twice a week for six weeks. The exercises will target both deep and superficial core muscles and focus on improving posture and body awareness. The program will include progressive adjustments to resistance and repetitions every two weeks.

Control Group: Participants in this group will receive educational sessions about proper posture and physical activity but will not engage in pilates exercises. They will have the option to participate in the pilates program after the study is completed.

B.Outcome Measures B.1. Trunk Endurance Extensor Endurance (Sorensen Test): Assesses the endurance of trunk extensor muscles by recording the duration the participant can hold a horizontal position against gravity.

Flexor Endurance Test: Measures the endurance of trunk flexor muscles by timing how long the participant can maintain a 60° flexion position.

B.2. Posture Analysis Postural alignment will be assessed using the Artificial Intelligence Posture Evaluation and Correction System (APECS) software, a photogrammetric tool for posture evaluation.

Markers will be placed on specific anatomical landmarks (e.g., ears, shoulders, hips, and knees) in static standing and sitting positions.

Photographs will be taken from the front, side, and back views to analyze:

Sagittal plane deviations (e.g., forward head posture, thoracic kyphosis). Frontal plane asymmetries (e.g., shoulder or pelvic tilts). Sitting posture deviations (e.g., cervical angle or slouched sitting positions).

Data will include angles and alignment deviations to quantify changes after the intervention.

B.3. Body Awareness Body Awareness Questionnaire (BAQ): Evaluates body awareness across physical, emotional, and social dimensions.

Objectified Body Consciousness Scale (OBCS): Measures dimensions of body monitoring, body shame, and appearance control beliefs.

C. Statistical Analysis Relationships between variables: Pearson's correlation coefficient will be used for normally distributed data, and Spearman's rank correlation will be applied for non-normally distributed data.

Between-group comparisons: The Independent Samples t-Test will be used for normally distributed data, and the Mann-Whitney U Test will be applied for non-parametric data.

Within-group comparisons: Paired t-Tests will be conducted for normally distributed data, and the Wilcoxon Signed Rank Test will be used for non-parametric data to assess changes from pre- to post-intervention.

Significance Level: All statistical analyses will be performed using the SPSS software package (version 26.0), with a significance level set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 10-19 years.
* Voluntary participation with signed informed consent.
* Ability to read and write in Turkish.

Exclusion Criteria:

* History of orthopedic injury within the last 3 months.
* Obesity (BMI > 30 kg/m²).
* Being under follow-up for a scoliosis diagnosis.

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-10-07 (Estimated); Study Completion 2025-10-07 (Estimated)

PRIMARY OUTCOMES:
Postural Alignment | Baseline and 6 weeks post-intervention.
  Evaluation of static postural alignment using the Artificial Intelligence Posture Evaluation and Correction System (APECS). Photos taken from front, side, and back will be analyzed to assess sagittal and frontal plane deviations, including cervical angle, shoulder alignment, and spinal curvature.
Trunk Endurance | Baseline and 6 weeks post-intervention.
  Assessment of core endurance using the Sorensen Test for trunk extensor muscles and the Flexor Endurance Test for trunk flexor muscles. The duration (in seconds) that participants can maintain the test position will be recorded.

SECONDARY OUTCOMES:
Objectified Body Consciousness Scale ( OBSC) | Baseline and 6 weeks post-intervention.
  Evaluation of body monitoring, body shame, and appearance control beliefs using the OBCS. Scores are calculated for each subscale individually.
Body Awareness Questionnaire (BAQ) | Baseline and 6 weeks post-intervention.
  Assessment of body awareness across emotional, physical, and social dimensions using the Body Awareness Questionnaire. Higher scores indicate better body awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Trakya University, Edirne, İskender, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No